CLINICAL TRIAL: NCT01716299
Title: Comparison of HIV Testing Algorithms in Two Sites in Ethiopia
Brief Title: Comparison of HIV Testing Algorithms
Status: Completed | Type: Observational
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Leslie Shanks, Medical Director, MSF-OCA, Medecins Sans Frontieres, Netherlands
Other Study IDs: msf09
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infection
Keywords: HIV; Diagnostics
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: application of a confirmation test — Addition of confirmation test to serial testing algorithm, including dilution test
Other: application of a confirmation test — use of rapid confirmation test

SUMMARY:
The primary objective of the study is to assess whether an improved MSF HIV diagnostic algorithm which includes a simple and easy to perform confirmation test has significantly better positive predictive value than WHO recommended RDT testing algorithms that do not include confirmatory testing.

DETAILED DESCRIPTION:
Rapid Diagnostic Tests (RDT's) are essential tools in antiretroviral treatment (ART) scale up. An important drawback to RDTs is the risk of false positive results. In 2005, MSF-Holland has therefore changed the testing algorithm to introduce a confirmation test. This proposal outlines an evaluation study of the results of the new confirmatory testing algorithm. It aims to compare the confirmatory algorithm employed by MSF-OCA to the MoH serial algorithm which is based on WHO recommendations. A secondary objective of the study is to determine if there is a correlation between kala-azar infection and risk of false positive HIV RDT results as clinicians in the projects suspect such a correlation. Furthermore, the study will look at the positive predictive value of weak test lines, which have been associated with higher risk of false positive results. Finally, the study aims to evaluate the results of a new simplified confirmation test, the dilution testing. Clients for the study will be recruited at two counseling and testing sites in Abdurafi and Humera, aiming to reach a sample size of 200 serial-algorithm positive and 200 negative samples in each site.

ELIGIBILITY:
Inclusion Criteria:

* • Age >= 59 months (to help ensure success of venepuncture)

  * Informed consent from the individual or guardian to participate in study

Exclusion Criteria:

* • Inability to obtain venous blood sample

  * Withdrawal of consent to test or to participate in the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting the Counseling and Testing centres in the two study sites
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
HIV result by Western Blot | one week

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Shanks, MD, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (2):
- Ethiopia (2):
  - Abdurafi Health Center, Ābderafī, Amhara Regional State
  - Humera Hospital, Humera, Tigray

REFERENCES:
- [Derived] Shanks L, Siddiqui MR, Abebe A, Piriou E, Pearce N, Ariti C, Masiga J, Muluneh L, Wazome J, Ritmeijer K, Klarkowski D. Dilution testing using rapid diagnostic tests in a HIV diagnostic algorithm: a novel alternative for confirmation testing in resource limited settings. Virol J. 2015 May 14;12:75. doi: 10.1186/s12985-015-0306-4. PMID 25972188
- [Derived] Shanks L, Siddiqui MR, Kliescikova J, Pearce N, Ariti C, Muluneh L, Pirou E, Ritmeijer K, Masiga J, Abebe A. Evaluation of HIV testing algorithms in Ethiopia: the role of the tie-breaker algorithm and weakly reacting test lines in contributing to a high rate of false positive HIV diagnoses. BMC Infect Dis. 2015 Feb 3;15:39. doi: 10.1186/s12879-015-0769-3. PMID 25645240